CLINICAL TRIAL: NCT00298116
Title: Molecular Associations With Reproductive Failure
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Crown Family Philanthropies (Other)
Responsible Party: Sponsor
Other Study IDs: 0502108
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Spontaneous Abortions; Infertility
MeSH Terms: conditions — Abortion, Spontaneous; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The overall hypothesis to be tested is: women with the molecular phenotype of highly skewed X chromosome inactivation are at increased risk of spontaneous abortion.

DETAILED DESCRIPTION:
The overall hypothesis to be tested is: women with the molecular phenotype of highly skewed X chromosome inactivation are at increased risk of spontaneous abortion.

We will investigate this hypothesis through two complimentary aims. In the Background and Significance section, we first present data on a 53-member pedigree segregating an X-linked recessive lethal defect that results in skewed X inactivation in the carrier females via secondary selection against those cells with the defective X chromosome active. We have characterized this deletion to be a 500 kb (approximate) deletion in distal Xq28. Moreover, the carrier females show a statistically significant increase in the frequency of spontaneous abortion as compared to non-deletion carrying relatives. Secondly, in the Preliminary Studies section, we present data from a population based case-control study wherein highly skewed X chromosome inactivation is significantly correlated with idiopathic recurrent spontaneous abortion. This protocol attempts to elucidate the mechanism underlying this association.

The first specific aim is to determine if women with highly skewed X chromosome inactivation are at risk of pregnancy loss. This will be accomplished through a prospective protocol, analyzing X chromosome inactivation patterns in pregnant women and investigating a possible association between X chromosome inactivation and pregnancy outcome. The second aim will study the nature of pregnancy loss in women with skewed X chromosome inactivation. This aim will correlate maternal X inactivation patterns with abortus karyotype.

ELIGIBILITY:
Inclusion Criteria:

* Patients are prospectively ascertained women with either a new pregnancy (specific aim 1), or a spontaneous abortion (specific aim 2).
* Given our enrollment strategy, we anticipate enrolling women between the ages of 18 and 45.

Exclusion Criteria:

* The study is limited only to females.
* Children are not eligible to participate in this study. Because the patient populations studied are (aim 1) women with primary infertility undergoing fertility treatment and (aim 2) women who have recently had a spontaneous abortion, the research topic is irrelevant to children.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients are recruited through Genetics during a counseling session.
Sampling Method: Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2000-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Skewed X-Inactivation is not associated with Reproductive Failure | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: W. Allen Hogge, MD, Principal Investigator — University of Pittsburgh and Magee-Womens Hospital
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States